CLINICAL TRIAL: NCT02173236
Title: The Effect of Platform Switching on Single Implants in the Esthetic Zone, Following Flapless Surgery and Early-Loading Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Yung-Ting Hsu, resident, Graduate Periodontics, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UM-
Record Dates: First submitted 2014-06-19; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: the Impact of Platform-switching
Keywords: Dental Implant Platform Switching; Early Dental Implant Loading

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- platform-switched implants (Experimental): platform-switched implants vs. platform-matched implants
  Interventions: Other: platform-matched implant
- platform-matched implants (Active Comparator): platform-switched implants vs. platform-matched implants
  Interventions: Other: platform-switched implants

INTERVENTIONS:
Other: platform-switched implants
  Other Names: SuperLine™, Dentium Inc., Cypress, CA
  Arms: platform-matched implants
Other: platform-matched implant
  Other Names: Zimmer TSV™, Zimmer Dental Inc., Carlsbad, CA
  Arms: platform-switched implants

SUMMARY:
The impact of platform switching with flapless surgery on early-loaded single-tooth implants on esthetic outcomes.

DETAILED DESCRIPTION:
Evaluation of clinical, radiographic and microbial outcomes of single implants with platform switching, compared to those with conventional platform.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be at least 18 years old and not currently pregnant
* Systemically healthy with no medical contraindications to implant surgery
* Having intact opposite tooth to proposed implant sites
* The edentulous ridge with minimal ridge deformities.

Exclusion Criteria:

* unstable medical status or conditions which may compromise wound healing
* osseous metabolic disorders (e.g., osteoporosis, Paget's disease etc.)
* uncontrolled dental or periodontal diseases
* edentulous ridges with the presence of fibrous dysplasia, severe tissue undercut, residual root, as well as insufficient dimensions or volume

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
plaque index | crown placement
  (Silness and Loe 1964). 0 represented the absence of plaque. 1 was the presence of plaque at gingival margin. 2 was the presence of visible plaque; whereas 3 was recorded if abundant plaque was observed
plaque index | post-loading 3 months
  (Silness and Loe 1964). 0 represented the absence of plaque. 1 was the presence of plaque at gingival margin. 2 was the presence of visible plaque; whereas 3 was recorded if abundant plaque was observed
plaque index | post-loading 6 months
  (Silness and Loe 1964). 0 represented the absence of plaque. 1 was the presence of plaque at gingival margin. 2 was the presence of visible plaque; whereas 3 was recorded if abundant plaque was observed
plaque index | post-loading 12 months
  (Silness and Loe 1964). 0 represented the absence of plaque. 1 was the presence of plaque at gingival margin. 2 was the presence of visible plaque; whereas 3 was recorded if abundant plaque was observed
gingival index | crown placement
  (Loe 1967) As for GI, normal gingival was scored as 0. 1 meant the presence of mild inflammation, slight change in color, slight edema and no BOP. Moderate inflammation was represented by 2, inclusive of the presence of gingival redness, edema, glazing and BOP. Severe inflammation with marked redness, edema, ulceration and spontaneous bleeding was scaled as 3
gingival index | post-loading 3 months
  As for GI, normal gingival was scored as 0. 1 meant the presence of mild inflammation, slight change in color, slight edema and no BOP. Moderate inflammation was represented by 2, inclusive of the presence of gingival redness, edema, glazing and BOP. Severe inflammation with marked redness, edema, ulceration and spontaneous bleeding was scaled as 3
gingival index | post-loading 6 months
  As for GI, normal gingival was scored as 0. 1 meant the presence of mild inflammation, slight change in color, slight edema and no BOP. Moderate inflammation was represented by 2, inclusive of the presence of gingival redness, edema, glazing and BOP. Severe inflammation with marked redness, edema, ulceration and spontaneous bleeding was scaled as 3
gingival index | post-loading 12 months
  As for GI, normal gingival was scored as 0. 1 meant the presence of mild inflammation, slight change in color, slight edema and no BOP. Moderate inflammation was represented by 2, inclusive of the presence of gingival redness, edema, glazing and BOP. Severe inflammation with marked redness, edema, ulceration and spontaneous bleeding was scaled as 3
Papillary index | crown placement
  (Jemt 1997) 0 = the absence of papilla, 1= <50% of the height of the gingival embrasure, 2= 50-99% of the height of the gingival embrasure, 3 = 100% of the proximal space, 4= overgrowth of the interproximal tissue
Papillary index | post-loading 3 months
  (Jemt 1997) 0 = the absence of papilla, 1= <50% of the height of the gingival embrasure, 2= 50-99% of the height of the gingival embrasure, 3 = 100% of the proximal space, 4= overgrowth of the interproximal tissue
Papillary index | post-loading 6 months
  (Jemt 1997) 0 = the absence of papilla, 1= <50% of the height of the gingival embrasure, 2= 50-99% of the height of the gingival embrasure, 3 = 100% of the proximal space, 4= overgrowth of the interproximal tissue
Papillary index | post-loading 12 months
  (Jemt 1997) 0 = the absence of papilla, 1= <50% of the height of the gingival embrasure, 2= 50-99% of the height of the gingival embrasure, 3 = 100% of the proximal space, 4= overgrowth of the interproximal tissue
The width of keratinized mucosa | crown placement
  measured at the midpoint on mid-facial surfaces of implants and adjacent two teeth.
The width of keratinized mucosa | post-loading 3 months
  measured at the midpoint on mid-facial surfaces of implants and adjacent two teeth.
The width of keratinized mucosa | post-loading 6 months
  measured at the midpoint on mid-facial surfaces of implants and adjacent two teeth.
The width of keratinized mucosa | post-loading 12 months
  measured at the midpoint on mid-facial surfaces of implants and adjacent two teeth.
Soft tissue level | crown placement
  the vertical distance from the gingival margin to the line connecting the facial gingival margin of two adjacent teeth
Soft tissue level | post-loading 3 months
  the vertical distance from the gingival margin to the line connecting the facial gingival margin of two adjacent teeth
Soft tissue level | post-loading 6 months
  the vertical distance from the gingival margin to the line connecting the facial gingival margin of two adjacent teeth
Soft tissue level | post-loading 12 months
  the vertical distance from the gingival margin to the line connecting the facial gingival margin of two adjacent teeth
Probing depth | crown placement
  Probing depth (PD) on the implant has also been recorded at 6 points mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual line-angles
Probing depth | post-loading 3 months
  Probing depth (PD) on the implant has also been recorded at 6 points mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual line-angles
Probing depth | post-loading 6 months
  Probing depth (PD) on the implant has also been recorded at 6 points mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual line-angles
Probing depth | post-loading 12 months
  Probing depth (PD) on the implant has also been recorded at 6 points mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual line-angles
marginal bone level changes | post-operative 2 weeks, immediately after crown delivery, 3, 6, and 12 months post-loading
  the vertical distance between alveolar crest to platform level (both mesial and distal)
ridge height | prior to surgery
  the distance from the highest point of alveolar crest to the base of the maxillary arch
ridge height | post-loading 12 months
  the distance from the highest point of alveolar crest to the base of the maxillary arch
ridge width 3mm below crest | prior to surgery
  the distance between the most prominent point on labial and palatal surfaces at the level of 3mm below the crest
ridge width 3mm below crest | post-loading 12 months
  the distance between the most prominent point on labial and palatal surfaces at the level of 3mm below the crest
ridge width 10 mm below crest | prior to surgery
  the distance between the most prominent point on labial and palatal surfaces at the level of 10 mm below the crest
ridge width 10 mm below crest | post-loading 12 months
  the distance between the most prominent point on labial and palatal surfaces at the level of 10 mm below the crest
the presence of perforation or dehiscence | post-loading 1 year
  using CBCT scan

SECONDARY OUTCOMES:
post-op experience | post-op 2weeks
  pain, bleeding, swelling and overall discomfort
microbial analysis | 12 months after loading
  peri-implant microbial profile
post-loading experience | post-op 12 months
  comfort, function (chewing/speaking), esthetics, and overall satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Graduate Periodontics, Department of Periodontics and Oral Medicine, University of Michigan School of Dentistry, Ann Arbor, Michigan, United States